CLINICAL TRIAL: NCT06840951
Title: Priming Cognitive Flexibility with RTMS to Enhance CBT for OCD: a Pilot Study
Brief Title: Priming CBT with RTMS for OCD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6236
Record Dates: First submitted 2025-02-07; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Obsessive compulsive disorder; Repetitive transcranial magnetic stimulation; Cognitive behavioural therapy; Flexibility; Neuroplasticity; Neurocognition
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Treatment-seeking participants at Sunnybrook Health Sciences Centre (SHSC) with a primary DSM-5 diagnosis of OCD (N = 10) will receive 10 sessions of rTMS followed by 12 weekly sessions of group CBT. All participants will complete repeated assessments at baseline, at the end of the rTMS (Session 10) treatment, and four times throughout the CBT treatment at weeks 1, 4, 8, and 12.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief rTMS + Group CBT (Experimental): Participants in this study arm will receive 10 sessions of rTMS treatment Monday through Friday for two weeks. Following rTMS treatment, participants will receive 12 weeks of CBT.
  Interventions: Device: rTMS; Behavioral: CBT
- Group CBT only (Active Comparator): Participants in this study arm will receive 12 weeks of CBT
  Interventions: Behavioral: CBT

INTERVENTIONS:
Device: rTMS — rTMS is a non-invasive procedure that uses electromagnetic field pulses to stimulate regions of the brain. rTMS can induce excitatory and inhibitory neural activity in the neural circuits of the motor cortex.
  Other Names: Repetitive transcranial magnetic stimulation
  Arms: Brief rTMS + Group CBT
Behavioral: CBT — CBT for OCD is a structured, short-term, present-oriented therapy with an emphasis on problem-solving and the modification of dysfunctional thinking and behaviour. CBT will be conducted in a group setting according to a session-by-session treatment manual that incorporates Exposure and Response Prevention (ERP) in the early phases of treatment and then increases emphasis on cognitive approaches for obsessions and compulsions with step-by-step strategies.
  Other Names: Cognitive behavioural therapy

SUMMARY:
Cognitive behavioural therapy (CBT), incorporating exposure/response prevention (ERP) and cognitive therapy, is considered the gold-standard first-line treatment for obsessive-compulsive disorder (OCD). Because CBT is a psychological treatment that aims to change patterns of thinking and behaving, it may be that improvement in cognitive functioning before treatment starts could lead CBT to be even more effective. One area of research that has shown potential benefit for OCD sufferers is rTMS. rTMS is a non-invasive procedure that uses pulses of energy to stimulate regions of the brain. Brief treatment with rTMS has shown to improve attention, memory, and other aspects of cognitive functioning that may facilitate learning in CBT. The proposed study aims to provide a pilot test of the clinical effectiveness of adding brief rTMS prior to completing CBT for OCD. If rTMS can demonstrate enhancement of cognitive functioning, which in turn, can improve treatment response to CBT, then the findings could easily be translated into routine clinical care.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) has a lifetime prevalence of close to three percent and is one of the leading causes of disability worldwide. In addition to being associated with significant functional impairment in daily living and quality of life, OCD has been associated with neurocognitive deficits. Meta-analyses have found that individuals with OCD tend to perform worse on measures of neurocognitive functioning, including aspects of memory and executive functioning, compared to healthy controls, and that symptom severity is associated with worse cognitive functioning. While effective treatments for symptoms of OCD have consistently been identified, research findings regarding the impact of these treatments on cognitive functions related to OCD have been mixed. In addition, cognitive behavioural therapy (CBT), which incorporates exposure/response prevention (ERP) and cognitive therapy, is considered the gold-standard treatment for OCD. However, a substantial proportion of clients fail to respond to the treatment, and the majority of treatment responders still continue to report impairing levels of symptoms. A possible novel therapeutic approach is the use of repetitive transcranial magnetic stimulation (rTMS), a non-invasive procedure that uses electromagnetic field pulses to stimulate regions of the brain. rTMS can induce excitatory and inhibitory neural activity in the neural circuits of the motor cortex. In OCD, rTMS has shown a moderate therapeutic effect on obsessive-compulsive disorder symptom severity with response rates surpassing those of sham conditions, and has shown to lead to significant improvements in cognitive functions such as working memory, executive functioning, and attention. There is emergent empirical literature supporting the synergistic effects of rTMS with CBT in a range of psychiatric conditions although this has yet to be tested directly in OCD.

The proposed study aims to provide a pilot, proof of principle test of the clinical efficacy and treatment mechanisms of adding brief rTMS prior to completing CBT for OCD for patient participants with DSM-5 diagnosed OCD. It also aims to provide a preliminary examination of the extent to which rTMS leads to neuropsychological improvement and the extent to which cognitive improvement relates to improved CBT treatment response. The primary goals are to compare the relative efficacy of rTMS plus CBT to CBT alone at reducing OCD symptoms, and to examine the extent to which neuropsychological change on measures of attention, memory, and executive functioning during rTMS relate to subsequent treatment success with CBT. Treatment outcomes will be assessed using standardized measures of OCD symptoms, as well as measures of mood, anxiety, and wellbeing. If this pilot study can demonstrate that a brief rTMS intervention of 10 sessions over a two-week period can confer significant clinical gains for those suffering with OCD through neuropsychological improvement and that these improvements, in turn, can enhance the effectiveness of CBT, then it could easily be translated into highly accessible, routine clinical care. Further, demonstration of improvement in OCD-associated neurophysiological dysfunction, given the refractory nature of the illness, would provide another avenue into the long-term enhancement of outcomes for this chronically affected population. Results will also add to our understanding of the role of psychological mechanisms in the pathogenesis and treatment response in OCD.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* experiencing clinically significant obsessive-compulsive symptoms based on the Yale-Brown Obsessive Compulsive Scale (YBOCS; score > 16)
* if on medications for OCD, must be stabilized, i.e., are currently receiving an adequate dose (equivalent of 40mg/day of fluoxetine) for an adequate duration (at least 8 weeks) prior to the initiation of the study

Exclusion Criteria:

* concurrent diagnosis of a severe mood disorder, schizophrenia or other psychotic disorders, or substance abuse/dependence
* suspected organic pathology
* an active comorbid medical condition that may require urgent intervention during the treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in OCD symptom severity (Yale-Brown Obsessive Compulsive Scale; Y-BOCS) | From baseline to post-CBT treatment, up to 19 weeks
  The Y-BOCS is a standardized rating scale measuring 10 items pertaining to obsessions and compulsions on a 5-point Likert scale ranging from 0 (no symptoms) to 4 (severe symptoms). Both the self-report and clinician interview versions of the Y-BOCS have been shown to possess high internal consistency and validity.

SECONDARY OUTCOMES:
Change in OCD symptom type (Obsessive Compulsive Inventory - Revised; OCI-R) | From baseline to post-CBT treatment, up to 19 weeks
  The OCI-R is a self -report short version of the OCI consisting of 18 items measuring six distinct factors: Washing, Checking, Ordering, Obsessing, Hoarding and Neutralizing. The items measuring Hoarding will not be analyzed based on the separation of OCD and hoarding disorder in the DSM-5. The OCI-R has been found to be a psychometrically sound and valid measure of OCD and its various symptom presentations.
Change in the experience of depression, anxiety, and stress symptoms (The Depression Anxiety Stress Scale - 21; DASS-21) | From baseline to post-CBT treatment, up to 19 weeks
  The DASS-21 is a self-report questionnaire comprising three subscales with seven items each for depression, anxiety and stress. The DASS-21 shows high internal consistency, high reliability in distinguishing between depression, anxiety and stress in adults, and good convergent and discriminant validity.
Change in various attitudes and beliefs related to obsessional thoughts (The Obsessional Beliefs Questionnaire; OBQ-44) | From baseline to post-CBT treatment, up to 19 weeks
  The OBQ-44 is a 44-item self-report questionnaire designed to assess the extent to which respondents agree or disagree with various attitudes and beliefs related to obsessional thoughts. The OBQ is internally consistent, and evidences good test-retest reliability, convergent validity, and discriminant validity.
Change in functional health and wellbeing (The Short Form 36-item Health Survey; SF-36) | From baseline to post-CBT treatment, up to 19 weeks
  The SF-36 Health Survey is a brief questionnaire containing 36 items about functional health and well-being. The reliability and validity of the SF-36 have been well documented. It has demonstrated good treatment sensitivity.
Change in the degree at which individuals find distress intolerable (The Distress Tolerance Scale; DTS) | From baseline to post-CBT treatment, up to 19 weeks
  The DTS is a 15-item self-report questionnaire that measures the degree to which individuals find distress intolerable, unacceptable, impairing, and necessary to avoid. The DTS has demonstrated strong psychometric properties.

OTHER OUTCOMES:
Change in performance of attention (CANTAB Motor Screening Task; MOT) | From baseline to post-rTMS treatment, 2 weeks
  The MOT evaluates potential sensorimotor or comprehension deficits.
Change in performance of sustained attention (CANTAB Rapid Visual Information Processing; RVP) | From baseline to post-rTMS treatment, 2 weeks
  The RVP measures sustained attention, latency, probability of false alarms, and sensitivity.
Change in performance of executive function (CANTAB One Touch Stockings of Cambridge; OTS) | From baseline to post-rTMS treatment, 2 weeks
  The OTS measures the working memory and spatial planning subdomains of executive function.
Change in performance of memory (CANTAB Verbal Recognition Memory task; VRM) | From baseline to post-rTMS treatment, 2 weeks
  The VRM measures new learning and verbal memory through the ability of collecting verbal information and its retrieval.
Change in performance of non-verbal memory (CANTAB Delayed Matching to Sample task; DMS) | From baseline to post-rTMS treatment, 2 weeks
  The DMS measures visual matching ability and short-term visual recognition memory.
Change in performance of non-verbal memory (CANTAB Paired Associates Learning task; PAL) | From baseline to post-rTMS treatment, 2 weeks
  The PAL measures visual memory and new learning.
Change in performance of social-emotional cognition (CANTAB Emotion Recognition Task; ERT) | From baseline to post-rTMS treatment, 2 weeks
  The ERT measures the ability in identification of six basic human emotions in facial expression along that expression's magnitude spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A. Rector, Ph.D., Principal Investigator — Sunnybrook Health Sciences Centre; Peter Giacobbe, M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada